CLINICAL TRIAL: NCT02860741
Title: Reducing Depressive Symptoms Among Rural African Americans
Acronym: REJOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 205181
Record Dates: First submitted 2016-08-05; First posted 2016-08-09 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Depressive Symptoms
Keywords: Sub-Clinical Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Churches in the REJOICE intervention arm will provide the REJOICE intervention over an 8 week period
  Interventions: Behavioral: REJOICE
- Control (Other): Churches in the control arm will receive an educational materials about both identifying depressive symptoms and managing depressive symptoms. This is consistent with self-management interventions commonly utilized for individuals experiencing subclinical levels of depressive symptoms.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: REJOICE — Small groups led by lay leaders undergo an 8-session faith-based behavioral activation protocol that provides individuals with education about: identifying depressive symptoms, identifying pleasurable activities, scheduling pleasurable activities, and identifying and addressing avoidant behaviors that act as barriers to completing pleasurable activities
  Arms: Intervention
Other: Control — Churches in the control arm will receive an educational materials about identifying depressive symptoms and self-management options for addressing depressive symptoms.
  Other Names: Usual Care
  Arms: Control

SUMMARY:
Rural African Americans are disproportionately impacted by social stressors that place them at risk for experiencing elevated depressive symptoms. This project will test the effectiveness of a culturally adapted behavioral activation intervention (REJOICE) for use within rural African American churches. Further, this project will gather data on strategies necessary to promote the successful implementation of this intervention within rural African American churches.

DETAILED DESCRIPTION:
Rural African Americans are disproportionately exposed to numerous stressors such as poverty, racism, and discrimination that place them at risk for experiencing elevated levels of depressive symptoms. Elevated levels of depressive symptoms can lead to a host of negative outcomes including both the development of and poor management of chronic illnesses (i.e. hypertension, diabetes, etc.), poor social functioning, poor occupational functioning, and development of clinical depression. Though effective treatments for decreasing depressive symptoms exist, rural African Americans often fail to receive adequate and timely care.

African American churches have been identified as potential venues for providing depression education and treatment for rural African Americans. Within the African American rural community, churches represent a key portal through which a large proportion (as much as 85%) of the African American community can be reached. Churches have been used to address physical health outcomes in those communities but few have focused primarily on addressing mental health outcomes.

Through the NIMHD funded project entitled, "Faith Academic Initiatives to Transform Health (FAITH) in the Delta", our partnership, consisting of faith community leaders and UAMS researchers, culturally adapted an evidence-based behavioral activation intervention for use with rural African American churches. This 8-session behavioral activation therapy was adapted to include faith-based themes, Scripture, and other aspects of the rural African American faith culture (e.g. bible studies, use of lay leaders to deliver the intervention). In addition to assessing the effectiveness of our intervention, ascertaining ways to implement this intervention with proper fidelity to maintain clinical outcomes is also critically important to increase the efficiency of translating research into practice. Work towards disseminating evidence-based depression interventions to "real world" settings is particularly salient in addressing depression disparities, whereby rural African Americans bear a disproportionate burden. Thus, this application proposes a Hybrid-2 pragmatic-effectiveness implementation trial that seeks to test the effectiveness of the culturally adapted evidence-based intervention and gather preliminary data on the strategies necessary to support successful implementation of this intervention in rural African American churches.

Specifically, this study aims to: 1) Refine a culturally appropriate, evidence-based depression intervention (REJOICE) based on results from our NIMHD-funded pilot study, 2) Determine whether REJOICE is superior to a usual-care control group at post treatment and a 3-month follow-up, 3) Collect pilot data regarding "real world" implementation strategies (i.e. face to face training and coaching calls) on the uptake and maintenance of REJOICE in rural African American churches.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Aged 18 and older
* Associated with a participating church through membership or participation in a church activity
* Free of medical problems that might contraindicate participation in a BA intervention (i.e. active intoxication (scores of 3 or more on the AUDIT-C), cognitive decline (score of 4 or more on the Brief Cognitive Screener51).

Exclusion Criteria:

* Individuals who are experiencing severe levels of depressive symptoms (scores of 21 or higher on BDI-II)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-05; Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms - Beck Depression Inventory (BDI-II) | Immediately upon completion of 8 week intervention
  The primary outcome of interest is evaluating differences in BDI-II scores among those individuals in the REJOICE cohort compared to those randomized into the control group during the T1 phase.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany F Haynes, PhD, Principal Investigator — Assistant Professor; Karen Yeary, PhD, Principal Investigator — Associate Professor; Camille Hart, MPH, Study Director — cnhart@uams.edu
Locations (4):
- United States (4):
  - Second Baptist Church of England, England, Arkansas
  - King Solomon, Helena, Arkansas
  - Greater Christ Temple, Little Rock, Arkansas
  - Evangelist Temple COGIC, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haynes T, Turner J, Smith J, Curran G, Bryant-Moore K, Ounpraseuth ST, Kramer T, Harris K, Hutchins E, Yeary KHK. Reducing depressive symptoms through behavioral activation in churches: A Hybrid-2 randomized effectiveness-implementation design. Contemp Clin Trials. 2018 Jan;64:22-29. doi: 10.1016/j.cct.2017.11.010. Epub 2017 Nov 21. PMID 29170075